CLINICAL TRIAL: NCT04273698
Title: What Can be Learnt From Offering Therapeutic Work to Parents and Infants (Under the Age of Five) in a Child and Adolescent Mental Health Service (CAMHS) Clinic That Does Not Routinely Offer This Type of Intervention?
Brief Title: What Can be Learnt From a Pilot Project Offering Brief Therapeutic Work to Parents and Infants in a Child and Adolescent Mental Health Service?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East London (Other)
Responsible Party: Principal Investigator, Rachel Allender, Chief investigator, University of East London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/SW/0020
Record Dates: First submitted 2020-02-13; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Infant Mental Health

STUDY DESIGN:
Intervention Model Description: Five families were each offered five parent-child psychotherapy sessions, based on the Tavistock Under-Fives model, and data was gathered and analysed from both the clinical intervention and from interviews and standardised outcome measures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical intervention (Experimental): The project involved recruiting families, with children under the age of five years old, who were experiencing one or more difficulties, and these families were offered five therapeutic sessions, based on a psychodynamic parent-infant psychotherapy approach.
  Interventions: Behavioral: Parent-infant psychotherapy

INTERVENTIONS:
Behavioral: Parent-infant psychotherapy — Brief psychoanalytic parent-infant psychotherapy

SUMMARY:
Can a method of working therapeutically with parents and children (under the age of five) be made use of in a Child and Adolescent Mental Health team, in which this kind of work does not regularly take place? I hope to understand whether this model of work can be helpful to the children and their families and to look at how this method was received by the team.

It is hoped that by working with the parents and child together, the families will be able to think about both the child's presenting difficulty, but also the relationship between the parents and their child and how the parents' own experiences and difficulties might impact on the present situation.

DETAILED DESCRIPTION:
The primary aim of this research is to trial an under-fives' service, in a Child and Adolescent Mental Health Service (CAMHS) team which has not offered this kind of work specifically before. The project would involve recruiting families, with children under the age of five years old, who are experiencing one or more difficulties, and these families would be offered five sessions, with the option of an additional five sessions, should this be required.

The work will broadly follow the Tavistock's model of parent-infant psychotherapy and the sessions will be centred within a psychodynamic psychotherapeutic framework. I hope that this trial will enable to me to learn more about this model of work, in terms of the processes involves and the themes that emerge. I hope to see how possible it is for this kind of work to be adopted within a generic CAMHS team, and how it is received by the families involved.

Due to this method of working being new to the team, it will be interesting to see how my colleagues respond to the model. It is likely that trying to gather full qualitative or quantitative data in this area would be beyond the scope of this piece of research, but I hope to make some reflections on how the model was received by the team. I hope to present the plan of work to the team prior to the treatment stage, and then share some of the findings from the research, after treatment. I also hope to conduct some form of consultation, with a staff group, following the treatment stage, in order to hear about their experiences of this method.

ELIGIBILITY:
Inclusion Criteria:

* The participants in this trial were children under the age of five years old, who had been referred to the CAMHS clinic.
* The child could have been experiencing a range of difficulties, including issues with sleeping, feeding or attachment, which were having an impact on their, or their families, functioning and wellbeing.
* The work involved working with the referred child and their parent(s) or carers

Exclusion Criteria:

* Families involved in court proceedings
* Families where there were safeguarding concerns
* Families currently experiencing domestic violence
* Families for whom severe parental mental health difficulties were indicated at the point of referral.
* Families who were already been accessing mental health support
* If the child had severe developmental difficulties and would require a specialist service
* Families requiring an interpreter in order to participate, I would have been unable to involve them, owing to the level of complexity this would have added in terms of the communication.

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
To learn how this method of therapeutic intervention was received by the families involved. The data gathered (in the form of process notes) from the interviews and therapy sessions was analysed using Thematic Analysis (Braun and Clarke, 2006). | 6 months
  The primary aim of this research was to trial an under-fives' service (like that developed at the Tavistock Clinic), in a CAMHS team which had not offered this kind of work specifically before, and to learn about the responses of families. The data gathered (in the form of process notes) from the interviews and therapy sessions was analysed using Thematic Analysis (Braun and Clarke, 2006).

SECONDARY OUTCOMES:
Goal Based Outcomes (GBO) measure | 6 months
  Each family was asked to set a goal which addressed the current problems or difficulties that they wanted to focus on during the therapy sessions. They were asked to rate their goal from zero to ten, zero representing that the goal is currently not being achieved at all, and ten meaning the goal has been entirely met. These goals were set at the start of treatment and reviewed and re-rated at the end.
Experience of Service questionnaire | 6 months
  At the end of the intervention, parents were also asked to complete an ESQ, which is a patient satisfaction measure, assessing their experience of the service, the intervention and clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lush, Study Director — Tavistock and Portman Trust
Locations (1):
- Shelley Clinic, CAMHS team, Dorset NHS, Bournemouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No